CLINICAL TRIAL: NCT04744454
Title: A Prospective, Single-arm, Open-label, Non-interventional, Multi-centre, Post Marketing Surveillance (PMS) Study of Cresemba to Evaluate Safety and Effectiveness in Patients With Invasive Aspergillosis or Invasive Mucormycosis in Korea
Brief Title: Post Marketing Surveillance (PMS) Study of Cresemba in Korea.
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C3791006; NCT04744454 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2020-12-16; First posted 2021-02-09 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Aspergillosis; Mucormycosis
Keywords: Aspergillosis; Mucormycosis; Isavuconazole; Korean
MeSH Terms: conditions — Aspergillosis; Mucormycosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Isauvuconazole group — Patients who are treated with Isavuconazole according to its protocol label.

SUMMARY:
The purpose of this study is to observe safety and effectiveness of Cresemba in patients with invasive Aspergillosis or invasive Mucormycosis in Korea during the post-marketing surveillance period as required by Ministry of Food and Drug Safety (MFDS).

DETAILED DESCRIPTION:
In compliance with the Korean New Drug Re-Examination Guidelines, this study aims to collect further observational data on the safety and effectiveness of Cresemba for six years after authorization is obtained in at least 600 subjects under routine clinical practice. As the safety and effectiveness results obtained from the clinical development program of Cresemba are based on randomized trials using specific inclusion and exclusion criteria, data from the present post-authorization study where Cresemba is used in routine clinical practice per approved label is anticipated to provide important information on safety and effectiveness in a real-world population in Korea. This non-interventional study is designated as a PMS study and is a commitment to MFDS.

ELIGIBILITY:
Inclusion Criteria: Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

* Patients aged 19 years or older
* Patients with proven or suspected diagnosis of invasive Aspergillosis or invasive Mucormycosis.
* Evidence of a signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria: Patients meeting any of the following criteria will not be included in the study:

* Patients with known hypersensitivity to the active substance of Isavuconazole or to any of the excipients.
* Patients are ineligible as determined by the investigator, such as those with familial short QT syndrome.
* Patients administrating ketoconazole, high-dose ritonavir (>200 mg every 12 hours) or strong CYP3A4/5 inducers (e.g. rifampicin, carbamazepine, phenytoin) that cannot be discontinued before administration of Cresemba.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is performed in accordance with routine clinical practice as per regulatory requirement. Therefore, inclusion and exclusion criteria relate to the labelled indication and contraindications. (Refer to the most updated version of the local product document [LPD]) All patients initiated on Isavuconazole and provided informed consent to the study will be enrolled continuously up to the planned number of enrolled patients. The assignment of the patient to Isavuconazole is decided by the investigator if he/she considers administering as per the current practice would provide clinical benefit with regards to safety and effectiveness.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Adverse event (AE) as safety evaluation | Starting from administration of first dose of Isavuconazole, will be continued through 28 days after from last administration of Isavuconazole.
  Incidence of the adverse events from baseline in all patients who received at least one dose of Isavuconazole and completed safety follow up will be assessed. AEs will be analyzed by preferred term coding.

SECONDARY OUTCOMES:
Effectiveness evaluation | From baseline to end of treatment or up to 12 weeks, whichever comes first.
  Effectiveness parameters- clinical response will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3791006